CLINICAL TRIAL: NCT00003692
Title: Video-Assisted Lobectomy for Peripheral (no Greater Than 3 cm), N0, Non-Small Cell Lung Cancer: A Phase II Feasibility Study
Brief Title: Video-Assisted Surgery in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39802; U10CA031946 (NIH); CLB-39802; E-C39802; CDR0000066795 (Registry Identifier: NCI Physicians Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
Keywords: occult non-small cell lung cancer; stage I non-small cell lung cancer; stage 0 non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Video-Assisted Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- video-assisted surgery (Experimental): Patients undergo video-assisted thoracic surgery (VATS) lobectomy, which requires 3 small incisions on the side of the chest. The entire anatomic pulmonary lobe is removed, as well as all peribronchial lymph nodes and anterior hilar lymph nodes. If it is not possible to remove the lobe using the VATS approach, then 1 of the incisions is converted to a standard thoracotomy. Patients are followed every 4 months for the first 2 years, and then every 6 months for the next 3 years.
  Interventions: Procedure: therapeutic thoracoscopy; Procedure: video-assisted surgery

INTERVENTIONS:
Procedure: therapeutic thoracoscopy
Procedure: video-assisted surgery

SUMMARY:
RATIONALE: Video-assisted surgery may be an effective treatment and have fewer side effects than conventional surgery in patients with non-small cell lung cancer.

PURPOSE: Phase II trial to study the effectiveness of video-assisted surgery in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of performing video-assisted thoracic surgery (VATS) lobectomy, without significant morbidity or perioperative mortality, in patients with small (no greater than 3.0 cm), peripheral, non-small cell lung cancer. II. Determine the rate at which a thoracotomy must be carried out to complete a VATS lobectomy in these patients. III. Describe the complications associated with this procedure. IV. Describe the length of the operative procedure, duration of chest tube stay, and length of hospitalization in this patient population. V. Describe the survival and failure-free survival, over a 5-year period, in this patient population following this procedure.

OUTLINE: Patients undergo video-assisted thoracic surgery (VATS) lobectomy, which requires 3 small incisions on the side of the chest. The entire anatomic pulmonary lobe is removed, as well as all peribronchial lymph nodes and anterior hilar lymph nodes. If it is not possible to remove the lobe using the VATS approach, then 1 of the incisions is converted to a standard thoracotomy. Patients are followed every 4 months for the first 2 years, and then every 6 months for the next 3 years.

PROJECTED ACCRUAL: A total of 135 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Suspected or histologically documented non-small cell lung cancer Solitary, peripheral lung lesion that is no greater than 3.0 cm No metastatic disease No positive lymph nodes at mediastinoscopy At least 5 years since diagnosis of non-small cell or small cell lung cancer

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: FEV1 at least 1.0 L or at least 50% of predicted Other: No significant comorbid medical or psychiatric condition No other active malignancy other than nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 1998-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
survival | up to 5 years
failure-free survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott J. Swanson, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center; John R. Roberts, MD, MBA, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (115):
- United States (112):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - University of California San Diego Cancer Center, La Jolla, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Swanson SJ, Herndon JE 2nd, D'Amico TA, Demmy TL, McKenna RJ Jr, Green MR, Sugarbaker DJ. Video-assisted thoracic surgery lobectomy: report of CALGB 39802--a prospective, multi-institution feasibility study. J Clin Oncol. 2007 Nov 1;25(31):4993-7. doi: 10.1200/JCO.2007.12.6649. PMID 17971599
- [Result] Swanson SJ, Herndon J, D'Amico A, et al.: Results of CALGB 39802: feasibility of video-assisted thoracic surgery (VATS) lobectomy for early stage lung cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1158, 2002.